CLINICAL TRIAL: NCT06931106
Title: Behavioral Intervention to Enhance HIV Pre-Exposure Prophylaxis Service Utilization Among Men Who Have Sex With Men in China Based on Health Action Process Approach and Conditional Economic Incentives
Brief Title: Behavioral Intervention for PrEP Service Utilization Among Chinese MSM: A HAPA and CEI Integrated Model
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Wangnan Cao, Associate Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00001052-24167
Record Dates: First submitted 2025-04-01; First posted 2025-04-17 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-04

CONDITIONS: HIV; PrEP; MSM; Behavior Changes
Keywords: HIV; pre-exposure prophylaxis; men who have sex with men; health action process approach; economic incentive
MeSH Terms: conditions — Homosexuality | interventions — Algenpantucel-L

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention group-B (Experimental): Participants will receive the AI-based HAPA and CEI behavioral intervention.
  Interventions: Behavioral: HAPA and CEI behavioral intervention
- Control group (No Intervention): Participants will receive non-personalized HIV prevention information, including free HIV testing and condom use, following the guidelines provided by the CDC and the operational standards of the community organizations, with weekly information push notifications.
- Intervention group-A (Experimental): Participants will receive HAPA-based behavioral intervention on the We-chat mini progarm.
  Interventions: Behavioral: HAPA-based intervention

INTERVENTIONS:
Behavioral: HAPA and CEI behavioral intervention — The intervention group will receive a 3-month technology-facilitated PrEP intervention and tailored messages will be developed using BCTs based on theoretical guidance. PrEP teleconsultations will be delivered by certified healthcare professionals, including infectious disease specialists, CDC-affiliated prevention officers, and MSM community leaders. Participants will be stratified into peer cohorts through algorithm-driven grouping based on demographic characteristics. Six participants will form a peer group, and the economic incentive amount will be based on the group-level PrEP initiation rates (verified by physician prescriptions). The economic incentive will decrease progressively based on the average completion rate within the group and will be divided into three tiers: 22 USD (completion rate of 80-100%), 11 USD (completion rate of 50-79%), and 0 USD (completion rate <50%).
  Arms: Intervention group-B
Behavioral: HAPA-based intervention — This group receives information pushes via a mini-program (3 messages per week) and two brief PrEP consultations; the first brief consultation is delivered jointly by community volunteers and a physician immediately after the baseline survey completion, based on a standardized consultation outline, and the second brief consultation is delivered jointly by community volunteers and a physician after the completion of the first monthly assessment (conducted within the mini-program), based on the standardized consultation outline and the results of that monthly assessment.
  Arms: Intervention group-A

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of a novel, intelligent intervention platform in bridging the "intention-behavior gap" for pre-exposure prophylaxis (PrEP) uptake among men who have sex with men (MSM) in China, a population at high risk for HIV infection. The study aims to address the following main questions:

* Can the intervention platform, guided by the Health Action Process Approach (HAPA) and Conditional Economic Incentive (CEI) dual-track theoretical framework, significantly increase PrEP initiation rates among MSM?
* What are the key mechanisms and pathways underlying the transition from PrEP intention to actual usage behavior?

Researchers will compare participants receiving the intelligent intervention platform (intervention group) with those receiving basic PrEP information (control group) to determine the platform's impact on PrEP initiation rates. Participants will:

* Use a mobile health platform equipped with personalized HIV risk assessments, PrEP knowledge resources, action planning tools, peer support features, and economic incentives.
* Complete baseline and follow-up surveys at 3 months and 6 months to assess PrEP initiation, adherence, and related behaviors.
* Engage in peer group activities and receive tailored feedback based on their progress.

This study seeks to provide evidence for scalable and sustainable strategies to improve PrEP uptake and contribute to HIV prevention efforts in high-risk populations.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years at enrollment;
* Assigned male at birth with a history of ≥1 male-male sexual encounter (anal or oral intercourse);
* HIV-negative confirmed by antibody testing at baseline;
* No prior use of PrEP;
* Expressed interest in PrEP intervention and commitment to complete scheduled follow-ups and data collection procedures;
* Mentally competent to provide informed consent and participate in decision-making;
* High HIV risk (meeting ≥1 of the following in the past 6 months): (1) Condomless anal/penile-vaginal intercourse; (2)Shared needle use during illicit drug injection; (3) Sexual contact with HIV-positive partner(s); (4) Newly diagnosed STI; (5) Repeated use of PEP for HIV prevention; or (6) Self-identified as PrEP candidate through voluntary request.

Exclusion Criteria:

* Confirmed HIV-positive status or unknown serostatus with refusal of HIV testing;
* Clinically significant health conditions contraindicating PrEP use (e.g., creatinine clearance <60 mL/min, documented hypersensitivity to PrEP components);
* Severe mental illness or neurological disorders impairing informed consent process.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
PrEP Initiation | 3 months
  The primary outcome indicators of this study is the rate of PrEP initiation, based on PrEP prescriptions issued by doctors.

SECONDARY OUTCOMES:
PrEP adherence | 3 months
  Secondary outcome indicators include the rate of PrEP adherence after initiating (based on self-reported adherence and the medication calendar in the program). Self-reported adherence: Assessed via validated questionnaires (e.g., visual analog scales or Likert scales) integrated into the mini-program, capturing missed doses, timing, and barriers. Medication calendar: Digitally tracked in the mini-program, recording daily PrEP intake with automated reminders and timestamped logs.
  Adherence rate calculated as the proportion of prescribed doses taken (e.g., ≥80% adherence threshold).
Intention to pay for PrEP | 3 months
  Structured questionnaires evaluating willingness to use three PrEP types (daily oral, on-demand, long-acting injectable) and maximum acceptable out-of-pocket payment (Likert scales (1-5) for willingness).
PrEP-related stigma | 3 months
  10-item HIV Pre-Exposure Prophylaxis Stigma Scale (HPSS) will be used to measure the PrEP-related stigma. The response format is 5-point Likert scale (1 = strongly disagree; 5 = strongly agree).
Changes in condomless sex | 3 months
  Retrospective self-reporting: Number of condomless acts in the past 3 months.
Changes in sexual partner numbers | 3 months
  Retrospective self-reporting: Number of sexual partners in the past 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Wangnan Cao, Ph.D, Principal Investigator — Peking University

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared publicly due to heightened privacy risks for MSM participants in China. Anonymization challenges and re-identification risks further limit safe sharing. Ethical approvals and informed consent agreements also restrict data use beyond the original study scope. Aggregated results will be published to ensure scientific transparency while safeguarding participant confidentiality.